CLINICAL TRIAL: NCT01972919
Title: MR Guided Phase II Radiotherapy Dose Escalation in Unresectable Non-metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Beth Erickson, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17687
Record Dates: First submitted 2013-08-29; First posted 2013-10-31 (Estimated); Results first posted 2025-02-10 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Unresectable Pancreatic Cancer
Keywords: Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiotherapy; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiation therapy plus chemotherapy (Experimental): MR guided dose escalated radiation therapy plus concurrent chemotherapy in unresectable non-metastatic pancreas cancer. Radiation therapy dose escalation to an MR-defined GTV of up to 69.75 Gy at 2.25 Gy per fraction and concurrent Gemcitabine or Capecitabine.
  Interventions: Radiation: Radiation Therapy; Drug: Concurrent chemotherapy (Gemcitabine, Capecitabine)

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation therapy dose escalation to an MR-defined gross tumor volume (GTV) of up to 69.75 Gy at 2.25 Gy per fraction.
  Other Names: Dose escalation radiation therapy
Drug: Concurrent chemotherapy (Gemcitabine, Capecitabine) — Gemcitabine 400mg/m^2 IV weekly x 6 doses. Capecitabine 825 mg/m^2 by mouth twice daily Monday-Friday on days of radiation use 500 mg tablets.
  Other Names: Gemzar; Xeloda

SUMMARY:
This research study is for people who have pancreas cancer for which surgery is not recommended. Potential patients must have already received several months of chemotherapy before they are eligible for this study and there will not have been any detectable spread of their tumor on imaging studies following this chemotherapy course.

DETAILED DESCRIPTION:
In this study the investigators want to find out more about the efficacy of giving higher doses of radiation with concurrent chemotherapy in controlling unresectable pancreas cancers than are used in either the pre-operative or post-operative setting. The investigators will assess acute and late side effects (problems and symptoms) of radiation therapy given at these higher doses of radiation (dose escalated) following full dose chemotherapy given before the radiation and with concurrent chemotherapy for pancreas cancer. Radiation therapy is given in higher doses that are limited by the proximity of normal organs to the radiation dose distribution to improve the likelihood of controlling the tumor in the pancreas while minimizing the risk of radiation injury to these organs. There are two chemotherapy drugs, Capecitabine is an oral drug taken twice per day on the same day that radiation therapy is given and Gemcitabine is an intravenous drug given once per week, during radiation therapy. Everyone in this study will have already received chemotherapy alone first. Everyone in this study will receive radiation therapy and concurrent chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed (histologic or cytologic), locally advanced, adenocarcinoma of the pancreas; patients must have unresectable disease based on institutional standardized criteria of unresectability or medical inoperability.
* Participants with and without regional adenopathy are eligible.
* No distant metastases, based upon the following minimum diagnostic workup:
* History/physical examination, including collection of weight and vital signs, within 28 days prior to study entry;
* Abdominal/pelvic CT scan with IV contrast within 21 days prior to study entry;
* Chest CT scan, or X-ray within 21 days prior to study entry.
* Abdominal/pelvic MR prior to radiation with perfusion and diffusion- weighted sequences and MR and CT sim for radiation planning Pet scan within 21 days prior to study entry, Functional renal study.
* Zubrod performance status 0-1 within 1 week of study entry.
* Age ≥ 18.
* Hematology and cancer antigen (CA) 19-9 / carcinoembryonic antigen (CEA) within 14 days prior to study entry, as follows.
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3;
* Platelets ≥ 100,000 cells/mm^3;
* Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.);
* Serum creatinine ≤ 1.5 mg/dl;
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 3 x upper limit of normal (ULN);
* Total bilirubin < 3.0 mg/dL;
* Alkaline phosphatase < 3 x ULN;
* Fasting blood glucose < 160 mg/dl.
* Negative serum pregnancy test (if applicable) within 14 days prior to study entry.
* Ability to swallow oral medications.
* Participants must have had at least 4 months of prior systemic chemotherapy.
* Participants must provide study specific informed consent prior to study entry.
* Women of childbearing potential and male participants who are sexually active must practice adequate contraception.

Exclusion criteria:

* Distant metastatic disease, second malignancy or peritoneal seeding;
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (For example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible).
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
* Any major surgery within 28 days prior to study entry
* Severe, active co-morbidity, defined as follows:
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
* Transmural myocardial infarction within 3 months prior to study entry;
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration;
* Uncontrolled malabsorption syndrome significantly affecting gastrointestinal function;
* Any unresolved bowel or bile duct obstruction;
* Major resection of the stomach or small bowel that could affect the absorption of capecitabine
* Acquired immune deficiency syndrome (AIDS) based upon current Center for Disease Control (CDC) definition;
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during the course of the study and for women, for 3 months after the last study drug administration.
* Women who are lactating at the time of registration and who plan to be lactating through 3 months after the last study drug administration.
* Prior allergic reaction to capecitabine or gemcitabine
* Inability to undergo an MR of the abdomen/pelvis
* Participation in another clinical treatment trial while on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-12-10 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2026-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Erickson, MD, Principal Investigator — Froedtert & The Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy Plus Chemotherapy: MR guided dose escalated radiation therapy plus concurrent chemotherapy in unresectable non-metastatic pancreas cancer. Radiation therapy dose escalation to an MR-defined GTV of up to 69.75 Gy at 2.25 Gy per fraction and concurrent Gemcitabine or Capecitabine.
  Radiation Therapy: Radiation therapy dose escalation to an MR-defined gross tumor volume (GTV) of up to 69.75 Gy at 2.25 Gy per fraction.
  Concurrent chemotherapy (Gemcitabine, Capecitabine): Gemcitabine 400mg/m^2 IV weekly x 6 doses.
  Capecitabine 825 mg/m^2 by mouth twice daily Monday-Friday on days of radiation use 500 mg tablets.
Period: Overall Study
Arm/Group | Radiation Therapy Plus Chemotherapy
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy Plus Chemotherapy
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: This measure will be the number of subjects alive at one and two years following the end of radiation treatment, up to two years and seven weeks.
Time Frame: 1 and 2 years following up to 7 weeks of radiation treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy Plus Chemotherapy
Number analyzed (Participants) | 23
Participants
  One Year | 13
  Two Years | 7

2. Secondary Outcome: Radiographic Response
Description: Number of participants treated with the proposed dose escalation achieving CR, PR, or SD measured by RECIST 1.1 criteria from magnetic resonance imaging (MRI), positron emission tomography (PET) or computed tomography (SC) scans.
Time Frame: Baseline and 1 year
Reporting Status: Not Posted

3. Secondary Outcome: Serum Cancer Antigen 19-9 (CA19-9)
Description: This measure will be the mean serum activity of CA19-9 in units/mL.
Time Frame: Baseline and 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Serum Carcinoembryonic Antigen (CEA)
Description: This measure will be the mean serum concentration of CEA in ng/mL.
Time Frame: Baseline and 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Radiation Induced Toxicity
Description: This measure will be the number of subjects experiencing a serious adverse event or grade three or higher non-serious adverse event by CTCAE v4.03 criteria that is definitely, likely, or possibly attributable to the radiation therapy.
Time Frame: 3 months post treatment
Reporting Status: Not Posted

6. Secondary Outcome: SMAD 4 Expression
Description: This measure will be the number of participants whose tumor biopsy is positive for the presence of SMAD 4 protein.
Time Frame: Baseline
Reporting Status: Not Posted

7. Secondary Outcome: Progression Free Survival
Description: This measure will be the number of subjects achieving a CR or PR or maintaining SD by RECIST 1.1 criteria one and two years following the end of radiation treatment.
Time Frame: 1 and 2 years
Reporting Status: Not Posted

8. Secondary Outcome: Efficacy of Dose Escalation
Description: This measure is the change from baseline of gross tumor volume for participants achieving a complete response (CR) or partial response (PR) or maintaining stable disease (SD) by RECIST 1.1 criteria.
Time Frame: Baseline and 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to two years and seven weeks.
Arm/Group | Radiation Therapy Plus Chemotherapy
All-Cause Mortality (participants affected / at risk) | 16/23
Serious Adverse Events (participants affected / at risk) | 4/23
Other Adverse Events (participants affected / at risk) | 10/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy Plus Chemotherapy (N=23)
Constipation (Gastrointestinal disorders) | 1 (1)
Bacteremia (Infections and infestations) | 2 (2)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy Plus Chemotherapy (N=23)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rotavirus (Gastrointestinal disorders) | 1 (1)
Gastric dysmotility (Gastrointestinal disorders) | 1 (1)
liver fibrosis (Gastrointestinal disorders) | 1 (1)
Portal Hypertension (Vascular disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Lymphocyte count decreased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/19/NCT01972919/Prot_SAP_000.pdf
  • Informed Consent Form (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT01972919/ICF_001.pdf